CLINICAL TRIAL: NCT02989701
Title: Pilot and Feasibility Trial of Plerixafor for Hematopoietic Stem Cell (HSC) Mobilization in Patients With Sickle Cell Disease
Brief Title: Pilot and Feasibility Trial of Plerixafor for Hematopoietic Stem Cell (HSC) Mobilization in Patients With Sickle Cell Disease Pilot and Feasibility Trial of Plerixafor for Hematopoietic Stem Cell (HSC) Mobilization in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alessandra Biffi (Other)
Responsible Party: Sponsor-Investigator, Alessandra Biffi, Director - Gene Therapy Program, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00023325
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Sickle Cell Disease Without Crisis
Keywords: Plerixafor
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Dose escalation of Plerixafor for Hematopoietic stem cell mobilization in patients with Sickle Cell Disease

SUMMARY:
Sickle cell disease (SCD) is one of the most common genetic diseases in the world. In North America, an estimated 2600 babies are born with SCD each year1, and approximately 70,000 to 100,000 individuals of all ages are affected in the United States2. The clinical manifestations of SCD include acute events, such as recurrent debilitating painful crises, as well as life-threatening pulmonary, cardiovascular, renal, and neurologic complications. The only established curative treatment for SCD patients is allogeneic hematopoietic stem cell transplant (HSCT). Unfortunately, access to this intervention is limited by availability of suitable matched donors, and HSCT is associated with significant morbidity and mortality. For patients who cannot undergo HSCT, treatment of SCD has been limited to one FDA-approved medication, hydroxyurea, and supportive symptomatic care. After decades with very few novel therapeutic options for SCD patients, autologous cell-based genetic therapies, including lentiviral-based gene therapy as well as gene editing, now offer the possibility of innovative curative approaches for patients lacking a matched donor for hematopoietic stem cell transplantation.

Gene therapy for sickle cell disease is increasingly promising, and there are currently open clinical trials at several centers that employ a gene addition strategy.

Options for autologous HSC collection include bone marrow harvest or peripheral blood HSC mobilization. Bone marrow (BM) harvest is an invasive procedure requiring anesthesia, which is associated with sickle cell-related morbidities, and may not achieve goal CD34+ cell dose, necessitating repeated procedures scheduled over multiple months. In most gene therapy trials, HSCs are obtained through peripheral collection after mobilization with granulocyte colony-stimulating factor (G-CSF) followed by peripheral blood (PB) apheresis. However, this approach is contraindicated in SCD because G-CSF has been reported to cause severe adverse effects in sickle cell patients. Even with doses sometimes smaller than standard, G-CSF has been shown to result in vaso-occlusive crises, severe acute chest syndrome, and in one report, massive splenomegaly and death. Alternative options for mobilization are needed.

Plerixafor has been compared to G-CSF in a sickle cell mouse model, and results showed effective mobilization of HSC subsets, without neutrophil or endothelial activation, and with lower total WBC and neutrophil counts compared to G-CSF-treated mice. Plerixafor use has not yet been documented in sickle cell patients. One other trial is currently open to test plerixafor in SCD patients (NCT02193191) but no results have yet been reported. Based on pre-clinical data, the mechanism of action of plerixafor, as well strategies the investigator will employ to mitigate risk, the investigator anticipates that it will be well-tolerated in the SCD patient population.

DETAILED DESCRIPTION:
This is a non-randomized pilot safety and feasibility single-center study which will treat subjects with SCD with plerixafor, followed by collection of peripheral HSPCs by apheresis. Accrual is a sample of up to 6 patients, with at least three patients treated with a plerixafor dose of 180 mcg/kg, and potential for escalation to a dose of 240 mcg/kg according to safety and tolerability of the lower dose. Three patients will be treated at the lower dose of 180 mcg/kg. If none of these patients experience a dose limiting toxicity (DLT), the next three patients will be treated with the higher dose of 240 mcg/kg. If one or more of the patients treated at 240 mcg/kg has a DLT, then 180 mcg/kg will be selected as the safe dose level. If no patients at the 240 mcg/kg have a DLT, then 240 mcg/kg will be selected as the safe dose level.

Within 30 days prior to plerixafor administration, subject will undergo laboratory testing, history, and physical exam. In order to retain the possibility for the subject to use his/her autologous cells for a future therapeutic indication, infectious disease testing and suitability for autologous transplant will be assessed per autologous transplant routine procedure.

If the subject is taking hydroxyurea, the medication will be stopped 14 days prior to the planned apheresis.

Between Days -7 and -2 prior to apheresis, the subject will undergo an exchange transfusion. This transfusion will be timed in accordance with the patient's existing chronic transfusion regimen. An exchange transfusion will be performed with post-transfusion hemoglobin electrophoresis confirming a %HbS of </= 30%.

After the exchange transfusion a bone marrow aspirate will be performed under local anesthesia or conscious sedation. The reason for performing the pre-plerixafor bone marrow is that in addition to our primary objective of assessing safety and feasibility of plerixafor in SCD patients, the investigator also aim to increase knowledge of HSPCs and their bone marrow niche in SCD patients - this will be relevant for better understanding basic disease pathophysiology, but also for the possible future use of BM HSPCs (obtained in basal conditions or after plerixafor administration) for gene therapy or gene editing therapies. It will be important to compare these phenotypic features in BM-derived cells versus plerixafor-derived cells. Additionally however, in order to also understand whether the HSPCs from SCD patients differ substantially from healthy donors, having a pre-plerixafor baseline sample of HSPCs from the same SCD subjects will provide important biological information as well.

On Day -1, the subject will be admitted to the Hematology service at Boston Children's Hospital. Confirmation of available, compatible units of packed red blood cells will be confirmed prior to administration of plerixafor (for use in case of an unexpected acute clinical need for transfusion). Labs will be drawn, including CBC, differential, hemoglobin electrophoresis, type and screen, and peripheral CD34+ cell count. The subject will receive a single dose of subcutaneous plerixafor.

On Day 0, prior to apheresis, labs will be drawn, including CBC, differential, and peripheral CD34+ count. Starting 6 hours after plerixafor dose, apheresis will be performed to collect 3-5x blood volumes. If the subject does not already have central venous access, access for apheresis will be obtained peripherally using 2 large bore 16g needles, and blood will be processed in the cell separator. Blood within the instrument will receive acid citrate dextrose formula A (ACD-A) (3%) at a rate of 1 mL/min/L of total blood volume, which is the standard apheresis dose. 2 grams of calcium gluconate is infused over the course of the procedure to prevent hypocalcemia associated with citrate administration. A CBC is drawn at the end of the procedure. Vital signs are monitored every 15 minutes while on the instrument. A second bone marrow aspirate will be performed before apheresis. The subject will remain admitted to the Hematology service overnight.

If excess cellular material is collected, a portion of the collected apheresis product (a minimum of 1 x 106 and a maximum of 3 x 106 unmanipulated CD34+ cells/kg) will be stored in clinically compliant conditions for any possible future use for the patient.

On Day + 1 after apheresis, labs will be drawn again including CBC, differential, and peripheral CD34+ count. The subject will be discharged from the Hematology service unless the subject does not meet standard clinical discharge criteria. On Day + 2 after apheresis, the study team will communicate with the subject via phone to inquire about any symptoms experienced. On Days +3, +7, +14, the subject will return for outpatient visit and labs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell disease with genotype HbSS, HbS/ Beta 0 thalassemia, HbSD, or HbSO.
2. Age 18-35 years.
3. Receiving regularly-scheduled blood transfusions as part of existing medical care.
4. Adequate hematologic parameters including:

   1. White blood cell (WBC) count within the range of 2.5 - 25.0 x 109 /L
   2. Hemoglobin within the range of 5 - 11 g/dL
   3. Platelet count within the range of 150 - 700 x 109 /L
5. Adequate organ function and performance status

   1. Karnofsky performance status ≥70%
   2. Serum creatinine </= 1.5 times the upper limit of normal for age, and calculated creatinine clearance or GFR >/= 60 mL/min/1.73 m2.
6. Patients who are taking hydroxyurea are allowed to be included in this study. Hydroxyurea will be stopped 14 days prior to planned day of apheresis.

Exclusion Criteria:

1. Patients who have uncontrolled illness including, but not limited to:

   1. Ongoing or active infection
   2. Emergency room admission or hospitalization for SCD-related reason in the past 30 days
   3. Major surgery in the past 30 days
   4. Medical/psychiatric illness/social situations that would limit compliance with study requirements as determined by the treating physician.
2. Known myelodysplasia of the bone marrow or abnormal bone marrow cytogenetics.
3. Receipt of an investigational study drug or procedure within 90 days of study enrollment.
4. Pregnant or breastfeeding.
5. Known acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on prior biopsy.
6. Known left ventricular ejection fraction <40% or known shortening fraction <25%.
7. Known DLCO (corrected for hemoglobin), FEV1, and/or FVC < 50% of predicted.
8. ALT > 2.5 X upper limit of normal or direct bilirubin > 2.0 mg/dL.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by monitoring for the occurrence of any described dose - limiting toxicities (DLTs) within 48 hours after dosing of plerixafor. | 14 days post dose
  Occurrence of death, ICU admission, stroke, vasoocclusive pain crisis (VOC) requiring continuous or scheduled parenteral opioid analgesia, acute chest syndrome, acute CNS event, or any other disease-related adverse event of grade 3 or higher.
Feasibility will be estimated by whether apheresis collection of a minimum of 0.5 X 106 CD34+ cells/kg is successful | 14 days post dose

SECONDARY OUTCOMES:
Pre-apheresis peripheral CD34+ cell concentration >/= 5 cells/µL. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Biffi, MD, Principal Investigator — Boston Children's Hospital; Erica Esrick, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States